CLINICAL TRIAL: NCT06885528
Title: UniCel DxH 900/690T Monocyte Distribution Width (MDW) Dual Cut-Off Clinical Accuracy Protocol
Brief Title: Adult MDW Dual Cut-Off Accuracy Study
Acronym: MDW
Status: Not yet recruiting | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Collaborators: Indiana University Health (Other); University of Kansas Medical Center (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: D25391
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Sepsis Diagnosis; MDW
MeSH Terms: conditions — Sepsis | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults presenting to Emergency Department: All-comers study of adults (18 to 89 years) of all races and ethnicities presenting to the Emergency Department
  Interventions: Diagnostic Test: Complete Blood Count with differential

INTERVENTIONS:
Diagnostic Test: Complete Blood Count with differential — First CBC w/diff test ordered within 12 hours of presentation to ED as part of standard medical care. The MDW result will be used as diagnostic marker to predict the risk of developing sepsis.

SUMMARY:
This study will establish the clinical performance of the Monocyte Distribution Width (MDW) parameter on the DxH 900/ DxH 690T hematology analyzers to aid in the detection and risk assessment of patients in the Emergency Department (ED) for progression to sepsis.

DETAILED DESCRIPTION:
The objective of this study is to validate the MDW dual cut-off values established during characterization and demonstrate the performance of MDW to detect sepsis in a multi-center study of adults presenting to the ED who have CBC w/diff ordered within 12 hours of presentation.

This study is designed to enroll all-comers from selected sites that currently have a DxH 900 in use as part of routine testing in the ED. All subjects who meet the Inclusion Criteria will be included in the study, without enrichment. Data from all subjects meeting the Inclusion Criteria will be provided to a panel of independent adjudicators. Adjudicators will be blinded to the MDW result and any sepsis diagnostic determinations which may or may not be in the original medical record.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 89 years) of all races and ethnicities presenting to the ED
* Whole Blood venous samples collected in K2EDTA while the patient was in the ED
* First CBC w/diff test ordered within 12 hours of presentation to ED as part of their standard medical care
* CBC w/diff tested within 2 hours of specimen collection
* Subjects with at least ≥12 hours of follow-up in the ED (or inpatient, if admitted) from presentation

Exclusion Criteria:

* CBC w/diff test ordered after 12 hours of presentation to ED
* Subjects previously enrolled in this study (i.e. subjects may not be enrolled more than once in this study)
* Subjects discharged from ED <12 hours from ED presentation
* ED Transfer Patients

Data Exclusions Post Enrollment:

* Samples that have a system generated flag from the Standard of Care (SOC) CBC w/diff testing will be excluded.
* Samples with instrument flags, including vote outs and review flags for MDW will also be excluded (i.e. invalid MDW results).
* Subjects' data collected with Instrument Quality Control failure(s).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers study of adult patients (18 to 89 years) of all races and ethnicities presenting to the ED
Sampling Method: Probability Sample
Enrollment: 2225 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of MDW | through study completion, an average of 1 year
  Clinical performance of MDW (expressed in terms of its interpretation bands and likelihood ratios) in diagnosing sepsis determined by clinical adjudication.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Drain, BSc, Study Director — Beckman Coulter, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; International Sepsis Definitions Conference. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Intensive Care Med. 2003 Apr;29(4):530-8. doi: 10.1007/s00134-003-1662-x. Epub 2003 Mar 28. PMID 12664219